CLINICAL TRIAL: NCT05994287
Title: Pain Treatment After Joint Surgery With a Combination of Aspirin, Ketorolac, and Celecoxib.
Brief Title: Pain Treatment With Combinations of NSAIDs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal State Budgetary Organization, Federal Center for Traumatology, Orthopedics and Arthroplasty (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2021-2
Record Dates: First submitted 2023-08-01; First posted 2023-08-16 (Actual); Last update posted 2024-01-25 (Actual); Status verified 2023-08

CONDITIONS: Postoperative Pain, Acute
Keywords: Postoperative pain; Non-steroidal anti-inflammatory drugs; Combination of NSAID; Aspirin; Ketorolac; Celecoxib
MeSH Terms: conditions — Pain, Postoperative | interventions — Aspirin; Ketorolac; Celecoxib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Drug: celecoxib (Active Comparator): The patients received celecoxib in a dose of 400 mg orally daily. The drug was prescribed from the second day of the operation for 5 days.
  Interventions: Drug: Celecoxib
- Drug: aspirin with ketorolac (Experimental): The patients received aspirin in a dose of 100 mg and ketorolac 90 mg orally daily. The drugs were prescribed from the second day of the operation for 5 days.
  Interventions: Drug: Aspirin; Drug: Ketorolac
- Drug: ketorolac and celecoxib (Experimental): The patients received ketorolac in a dose of 90 mg and celecoxib 400 mg orally daily. The drugs were prescribed from the second day of the operation for 5 days.
  Interventions: Drug: Ketorolac; Drug: Celecoxib
- Drug: aspirin, ketorolac and celecoxib (Active Comparator): The patients received aspirin in a dose of 200 mg, ketorolac 90 mg, and celecoxib 400 mg orally daily. The drugs were prescribed from the second day of the operation for 5 days.
  Interventions: Drug: Aspirin; Drug: Ketorolac; Drug: Celecoxib

INTERVENTIONS:
Drug: Aspirin — The patients received aspirin in a dose of 100 mg orally daily.
  Arms: Drug: aspirin with ketorolac; Drug: aspirin, ketorolac and celecoxib
Drug: Ketorolac — The patients received ketorolac in a dose of 90 mg mg orally daily.
  Arms: Drug: aspirin with ketorolac; Drug: aspirin, ketorolac and celecoxib; Drug: ketorolac and celecoxib
Drug: Celecoxib — The patients received celecoxib in a dose of 400 mg orally daily.
  Arms: Drug: aspirin, ketorolac and celecoxib; Drug: celecoxib; Drug: ketorolac and celecoxib

SUMMARY:
The search for new safe and effective methods of pain relief after surgery on large joints is still an urgent problem. The most optimal approach in the treatment of postoperative pain is the use of multimodal analgesia with a different mechanism of action that act on various mechanisms of pain and can include opioids, nonsteroidal anti-inflammatory drugs (NSAIDs), acetaminophen, anticonvulsants, NMDA antagonists, alpha-2-agonists, and sodium and calcium channel blocking agents, as well as local anesthetics. NSAIDs are the most popular and safe means for pain relief. Therefore, a lot of efforts are aimed at increasing the effectiveness of NSAIDs use. The aim of this study was to evaluate the effectiveness of simultaneously administering two or three NSAIDs, compared to using only one NSAID, for pain relief after surgery on large joints such as hip or knee arthroplasty.

DETAILED DESCRIPTION:
This is 6 days, randomized, double blind, parallel group, single-center study in 105 subjects. The distribution into groups was carried out by sequentially alternating the set into 4 groups celecoxib 400 mg orally daily, aspirin 100 mg and ketorolac 90 mg orally daily, ketorolac 90 mg and celecoxib 400 mg orally daily; aspirin 200 mg, ketorolac 90 mg and celecoxib 400 mg orally daily.

ELIGIBILITY:
Inclusion Criteria:

* The patients with diagnosis of osteoarthritis of the knee or hip joint (M15.0, M16, M17) after primary knee or hip arthroplasty.
* Informed consent.

Exclusion Criteria:

* Patients who cannot cooperate with the trial.
* Pregnant or breast feeding women,
* Оpioid addiction,
* Contraindication to NSAIDs (allergy to NSAID, history of ulcer and gastrointestinal bleeding, liver failure, renal failure (eGRF < 60 ml/kg/1,73m2) and chronic kidney disease 2-5, known thrombocytopenia (<100 mia/L)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2022-01-01 (Actual); Study Completion 2023-01-01 (Actual)

PRIMARY OUTCOMES:
Measuring postoperative pain using the visual analog scale for pain (VAS-P) | 5 days
  The patients choose the score on the 10 cm line scale with (VAS-P) rage from 0 ('no pain') to 10 (severe pain).

SECONDARY OUTCOMES:
Arachidonic acid-stimulated platelet tests | 5 days
  Assessed by Multiplate ASPItest, Roche Diagnostics GmbH. The platelet aggregation expressed in arbitrary aggregation units (AU) multiplied by the recorded time in minutes (AU*min).
Hemoglobin | 5 days
  Hemoglobin (HGB) level in g/L
Hematocrit | 5 days
  Hematocrit level in %
Erythrocytes | 5 days
  Erythrocytes (RBC) number in 1 litter
Platelets cells | 5 days
  Platelets cells (PLT) number in 1 litter
Fibrinogen | 5 days
  Fibrinogen level in g/L
Partial thromboplastin time | 5 days
  Partial thromboplastin time (PTT) in seconds
Prothrombin time | 5 days
  Prothrombin time in %

CONTACTS AND LOCATIONS:
Overall Officials: Vladimir U. Emelianov, MD PhD, Principal Investigator — Federal Center for Traumatology, Orthopedics and Arthroplasty, Cheboksary, Russia
Locations (1):
- Federal Center for Traumatology, Orthopedics and Endoprosthetics, Cheboksary, Chuvashskaya Respublika, Russia